CLINICAL TRIAL: NCT04150666
Title: The Water Intake Trail and Primary Aldosteronism Postoperation(WIT-PAP)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects are willing to participating.
Sponsor: Qifu Li (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary Investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WIT-PAP Study 2019
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Hyperaldosteronism; Renal Insufficiency
Keywords: primary aldosteronism; surgery therapy; water intake; renal function
MeSH Terms: conditions — Hyperaldosteronism; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydration (Experimental): Participants randomized to the hydration-intervention group will be asked to drink 2.0 to 2.5 L of water per day (depending on sex), in addition to usual consumed beverages, for 3 months
  Interventions: Dietary Supplement: Hydration
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Hydration — the same with arm descriptions
  Arms: Hydration

SUMMARY:
To investigate whether increasing water intake has renal protective effect on PA patients after surgical treatment.

DETAILED DESCRIPTION:
This is a single-center randomized controlled trial study to verify the effect of drinking water on renal function after PA surgery treatment and to follow up the clinical outcomes. We will take short-term follow-up on whether increasing water intake can improve eGFR decline in the early stage of PA patients after surgical treatment and further long-term follow-up to investigate whether increasing drinking water has long-term memory effect to slow down renal function deterioration and improve clinical outcomes. This study will be completed in 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Able to provide informed consent and willing to complete follow-up visits.
* Estimated glomerular filtration(eGFR) rate over 60 ml/min/1•73 m²
* According to the Guideline of Primary Aldosteronism, unilateral PA has been diagnosed and unilateral adrenalectomy has been completed
* Urine volume can be recorded consciously, and daily drinking water volume is less than 2L/d

Exclusion Criteria:

* Pregnant or breastfeeding
* Diagnosed with other types of chronic kidney diseases, such as IgA nephropathy, lupus nephritis, etc.
* History of malignant tumor
* History of kidney stones in past 5 years
* Kidney transplant within past six months (or on waiting list)
* Less than two years life expectancy
* Serum sodium <130 mEq/L without suitable explanation or Serum calcium >2.6 mmol/L without suitable explanation
* Currently taking hydrochlorothiazide >25 mg/d, indapamide >1.25 mg/d, furosemide >40 mg, or metolazone >2.5 mg/d
* Poor blood pressure control (systolic pressure>180mmHg or diastolic pressure> 110mmHg)
* Alcoholics, drug addicts, and people with mental disorders who cannot cooperate
* Patient is under fluid restriction (<1.5 L a day) for kidney disease, heart failure, or liver disease, AND meets any of the following criteria: i) end stage of the disease (heart left ventricular ejection fraction <40%, NYHA class 3 or 4, or end stage cirrhosis) , ii) hospitalization secondary to ACS,heart failure, stroke,ascites and/or anasarca ,iii)Severe anemia (Hb<60g/L)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Renal decline | Baseline and 3 months
  Change in estimated glomerular filtration rate between baseline and 3 months

SECONDARY OUTCOMES:
24-hour urine albumin | Baseline,3 and 6 months
  Change in 24-hour urine albumin among baseline, 3 and 6 months
Rapid renal decline | Baseline 3, and 6 months
  Proportion with eGFR (estimated glomerular filtration rate) decline >5% among Baseline 3, and 6 months
Measured creatinine clearance | Baseline 3, and 6 months
  Change in measured creatinine clearance among baseline, 3 and 6 months
Copeptin | Baseline 3, and 6 months
  Change in copeptin among baseline, 3 and 6 months
Blood pressure | Baseline 3, and 6 months
  Change in blood pressure among baseline, 3 and 6 months
Waist circumference | Baseline 3, and 6 months
  Change in waist circumference among baseline, 3 and 6 months
Body mass index | Baseline 3, and 6 months
  Change in body mass index among baseline, 3 and 6 months
Renal events | Baseline and 12 months
  Two of the three morning urine UACR&>300 mg/g Cr, or 24-hour urine protein >300 mg/ 24 h, or serum creatinine level doubled and reached at least 200 μmol/l(2.26 mg/dl), or required renal replacement therapy, or died of renal diseases

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nishikawa T, Omura M, Saito J, Matsuzawa Y, Kino T. Editorial comment from Dr Nishikawa et al. to preoperative masked renal damage in japanese patients with primary aldosteronism: identification of predictors for chronic kidney disease manifested after adrenalectomy. Int J Urol. 2013 Jul;20(7):693-4. doi: 10.1111/iju.12052. Epub 2012 Dec 11. No abstract available. PMID 23231595
- [Result] Nakano Y, Yoshimoto T, Fukuda T, Murakami M, Bouchi R, Minami I, Hashimoto K, Fujii Y, Kihara K, Ogawa Y. Effect of Eplerenone on the Glomerular Filtration Rate (GFR) in Primary Aldosteronism: Sequential Changes in the GFR During Preoperative Eplerenone Treatment to Subsequent Adrenalectomy. Intern Med. 2018 Sep 1;57(17):2459-2466. doi: 10.2169/internalmedicine.0438-17. Epub 2018 Apr 27. PMID 29709927
- [Result] Hundemer GL, Curhan GC, Yozamp N, Wang M, Vaidya A. Renal Outcomes in Medically and Surgically Treated Primary Aldosteronism. Hypertension. 2018 Sep;72(3):658-666. doi: 10.1161/HYPERTENSIONAHA.118.11568. PMID 29987110
- [Result] Clark WF, Sontrop JM, Huang SH, Gallo K, Moist L, House AA, Cuerden MS, Weir MA, Bagga A, Brimble S, Burke A, Muirhead N, Pandeya S, Garg AX. Effect of Coaching to Increase Water Intake on Kidney Function Decline in Adults With Chronic Kidney Disease: The CKD WIT Randomized Clinical Trial. JAMA. 2018 May 8;319(18):1870-1879. doi: 10.1001/jama.2018.4930. PMID 29801012